CLINICAL TRIAL: NCT00360295
Title: A Multicenter, Non-Randomized, Open Label Trial Of Azithromycin SR For The Treatment Of Mild To Moderate Community Acquired Pneumonia In Japanese Adults
Brief Title: A Trial Of Azithromycin SR For The Treatment Of Mild To Moderate Community Acquired Pneumonia In Japanese Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0661174
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Pneumonia, Community-Acquired
MeSH Terms: conditions — Community-Acquired Pneumonia

INTERVENTIONS:
Drug: Azithromycin SR

SUMMARY:
To evaluate the clinical efficacy and safety in patients with mild or moderate community-acquired pneumonia receiving a dose of 2 g of azithromycin in the SR formulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as mild or moderate in severity by the classification of pneumonia "Clinical evaluation methods for new antimicrobial agents to treat respiratory infections: Report of the Committee for the Respiratory System, Japan Society of Chemotherapy (established in 2000)".

Exclusion Criteria:

* Severe underlying disease; patients in which drug clinical evaluation is difficult because of confounding diseases. ("Severe" assessed by the Severity of underlying diseases and complications of "Clinical evaluation methods for new antimicrobial agents to treat respiratory infections (draft)" by the Japan Society of Chemotherapy (1997)).

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2006-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is Data Review Committee's Clinical efficacy at Day 8.

SECONDARY OUTCOMES:
Data Review Committee's clinical efficacy (at Day 15 and 29) Investigator's clinical efficacy (at Day 8, 15 and 29), and the tendency toward clinical improvement (at Day 4) Bacteriological efficacy (at Day 4, 8, 15 and 29)
Adverse events and safety Laboratory data

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- Japan (46):
  - Pfizer Investigational Site, Asahi, Chiba
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Higashi, Fukuoka
  - Pfizer Investigational Site, Kasuya-gun, Fukuoka
  - Pfizer Investigational Site, Munakata, Fukuoka
  - Pfizer Investigational Site, Nishiku, Fukuoka
  - Pfizer Investigational Site, Isesaki, Gunma
  - Pfizer Investigational Site, Maebashi, Gunma
  - Pfizer Investigational Site, Asahikawa, Hokkaido
  - Pfizer Investigational Site, Kamikawa-gun, Hokkaido
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Teine, Hokkaido
  - Pfizer Investigational Site, Hitachi, Ibaraki
  - Pfizer Investigational Site, Hitachi-Naka, Ibaraki
  - Pfizer Investigational Site, Kasama, Ibaraki
  - Pfizer Investigational Site, Moriya, Ibaraki
  - Pfizer Investigational Site, Toride, Ibaraki
  - Pfizer Investigational Site, Tsuchiura, Ibaraki
  - Pfizer Investigational Site, Marugame, Kagawa-ken
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Yokosuka, Kangawa
  - Pfizer Investigational Site, Emukae, Kitamatsuura, Nagasaki
  - Pfizer Investigational Site, Hirase-cho, Sasebo,, Nagasaki
  - Pfizer Investigational Site, Nagasaki, Nagasaki
  - Pfizer Investigational Site, Shigesato-cho, Nagasaki, Nagasaki
  - Pfizer Investigational Site, Ohte-machi, Oita City, Oita Prefecture
  - Pfizer Investigational Site, Oita City, Oita, Oita Prefecture
  - Pfizer Investigational Site, Ōita, Oita Prefecture
  - Pfizer Investigational Site, Tanaka-machi, Oita, Oita Prefecture
  - Pfizer Investigational Site, Yufu, Oita Prefecture
  - Pfizer Investigational Site, Naha, Okinawa
  - Pfizer Investigational Site, Nakagami-gun, Okinawa
  - Pfizer Investigational Site, Okinawa, Okinawa
  - Pfizer Investigational Site, Shimajiri-gun, Okinawa
  - Pfizer Investigational Site, Daitō, Osaka
  - Pfizer Investigational Site, Katano, Osaka
  - Pfizer Investigational Site, Kita-ku, Osaka
  - Pfizer Investigational Site, Koshigaya, Saitama
  - Pfizer Investigational Site, Kiyose, Tokyo
  - Pfizer Investigational Site, Nakano City, Tokyo
  - Pfizer Investigational Site, Ōme, Tokyo
  - Pfizer Investigational Site, Setagaya City, Tokyo
  - Pfizer Investigational Site, Shinagawa, Tokyo
  - Pfizer Investigational Site, Sumida City, Tokyo
  - Pfizer Investigational Site, Yamagata, Yamagata
  - Pfizer Investigational Site, Yonezawa, Yamagata

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661174&StudyName=A%20Trial%20Of%20Azithromycin%20SR%20For%20The%20Treatment%20Of%20Mild%20To%20Moderate%20Community%20Acquired%20Pneumonia%20In%20Japan%20Adults